CLINICAL TRIAL: NCT03783559
Title: TACE Associated With Systemic Chemotherapy Versus Systemic Chemotherapy in Patients Who Failed With First Line Chemotherapy
Brief Title: TACE(Transcatheter Arterial Chemoembolization ) Associated With Systemic Chemotherapy Versus Systemic Chemotherapy Alone in Patients With Unresectable CRLM(Colorectal Liver Metastases)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACECRLM
Record Dates: First submitted 2018-12-15; First posted 2018-12-21 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Adenocarcinoma Metastatic to the Liver
Keywords: colorectal cancer liver metastasis; Transarterial chemoembolization; conversion resection rates; chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): TACE plus chemotherapy ± target therapy
  Interventions: Drug: TACE; Drug: chemotherapy±target therapy
- Arm B (Active Comparator): chemotherapy ± target therapy
  Interventions: Drug: chemotherapy±target therapy

INTERVENTIONS:
Drug: TACE — TACE
  Arms: Arm A
Drug: chemotherapy±target therapy — chemotherapy±target therapy

SUMMARY:
To date no randomized controlled trials have been completed that demonstrated whether TACE(Transarterial chemoembolization) is an effective adjunct to systemic chemotherapy (target therapy) with respect to advantages in conversion resection rates and survival compared with chemotherapy (target therapy) alone for patients who failed with first-line chemotherapy.The primary objective of this trial is to determine conversion resection rates and survival for patients with colorectal cancer liver metastasis are treated with TACE plus chemotherapy ± target therapy, compared to chemotherapy ± target therapy in the 2nd, and 3rd line.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed CRLM
* disease limited to the liver Unresectable disease by surgery or other local therapies
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2,child pugh A or B
* Expected survival ≥ 3 months
* Adequate hematological, hepatic and renal function
* PD(progressive disease) after first line chemotherapy

Exclusion Criteria:

* pregnant or lactating women
* patients with severe organ dysfunction or failure
* with severe cardiovascular or mental disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 months

SECONDARY OUTCOMES:
overall survival | 6 months
conversion resection rates | 2-4months

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, PhD, Study Chair — Fudan University
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Liu Y, Chang W, Zhou B, Wei Y, Tang W, Liang F, Chen Y, Yan Z, Lv M, Ren L, Xu J. Conventional transarterial chemoembolization combined with systemic therapy versus systemic therapy alone as second-line treatment for unresectable colorectal liver metastases: randomized clinical trial. Br J Surg. 2021 Apr 30;108(4):373-379. doi: 10.1093/bjs/znaa155. PMID 33611431
- [Derived] Swierz MJ, Storman D, Riemsma RP, Wolff R, Mitus JW, Pedziwiatr M, Kleijnen J, Bala MM. Transarterial (chemo)embolisation versus no intervention or placebo for liver metastases. Cochrane Database Syst Rev. 2020 Mar 12;3(3):CD009498. doi: 10.1002/14651858.CD009498.pub4. PMID 32163181